CLINICAL TRIAL: NCT05216341
Title: A 2-stage, Phase 2a Study to Evaluate the Efficacy, Safety, and Tolerability of OLP-1002 Subcutaneous Injections for Reducing Moderate to Severe Pain Due to Osteoarthritis in a Hip and/or Knee Joint
Brief Title: Study of OLP-1002 Injections for Reducing Moderate to Severe Pain Due to Osteoarthritis in Hip and/or Knee Joint
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OliPass Corporation (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OLP-1002-002A
Record Dates: First submitted 2021-12-20; First posted 2022-01-31 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: Stage 1 - open label, dose-finding study, single ascending dose design
  Stage 2 - double-blind, placebo-controlled, parallel-arm study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stage 1: open label
  Stage 2: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Stage 1: Arm 1 (OLP-1002, 1 μg) (Experimental): Participants will receive once single dose of 1 μg OLP-1002 on Day 1
  Mode of Administration: subcutaneously injection
  Interventions: Drug: OLP-1002
- Stage 1: Arm 2 (OLP-1002, 3 μg) (Experimental): Participants will receive once single dose of 3 μg OLP-1002 on Day 1
  Mode of Administration: subcutaneously injection
  Interventions: Drug: OLP-1002
- Stage 1: Arm 3 (OLP-1002, 10 μg) (Experimental): Participants will receive once single dose of 10 μg OLP-1002 on Day 1
  Mode of Administration: subcutaneously injection
  Interventions: Drug: OLP-1002
- Stage 1: Arm 4 (OLP-1002, 25 μg) (Experimental): Participants will receive once single dose of 25 μg OLP-1002 on Day 1
  Mode of Administration: subcutaneously injection
  Interventions: Drug: OLP-1002
- Stage 1: Arm 5 (OLP-1002, 50 μg) (Experimental): Participants will receive once single dose of 50 μg OLP-1002 on Day 1
  Mode of Administration: subcutaneously injection
  Interventions: Drug: OLP-1002
- Stage 1: Arm 6 (OLP-1002, 80 μg) (Experimental): Participants will receive once single dose of 80 μg OLP-1002 on Day 1
  Mode of Administration: subcutaneously injection
  Interventions: Drug: OLP-1002
- Stage 2: Arm 1 (OLP-1002, 1μg) (Experimental): Participants will be randomised to receive single dose of 1μg OLP-1002 on Day 1
  Mode of Administration: subcutaneously injection
  Interventions: Drug: OLP-1002
- Stage 2: Arm 2 (OLP-1002, 2μg) (Experimental): Participants will be randomised to receive single dose of 2μg OLP-1002 on Day 1
  Mode of Administration: subcutaneously injection
  Interventions: Drug: OLP-1002
- Stage 2: Arm 3 (Placebo) (Placebo Comparator): Participants will be randomised to receive single dose of Placebo on Day 1
  Mode of Administration: subcutaneously injection
  Interventions: Drug: OLP-1002

INTERVENTIONS:
Drug: OLP-1002 — Stage 1: A total of 5 participants will be enrolled in each arm in Stage 1.
  Each participant will receive one single dose of OLP-1002 by subcutaneous injection.
  Stage 2: Up to 90 participants will be randomised on Day 1 to one of 3 treatment arms, in the ratio of 1:1:1 to receive one single dose of OLP-1002 (1 µg or 2 µg) or placebo.
  Each participant will receive one single dose of OLP-1002 or placebo by subcutaneous injection.
  Other Names: Diluent (Placebo) - Only for Stage 2

SUMMARY:
The study is designed to evaluate the efficacy, safety and tolerability of OLP-1002 Subcutaneous (SC) injections for reducing moderate to severe pain due to osteoarthritis in a hip and/or knee joint.

DETAILED DESCRIPTION:
The study consists of two Stages (Stage 1 and Stage 2)

Stage 1: It is an open-label, dose-finding study employing a single ascending dose design to determine appropriate dose level starting dose of OLP-1002 for Stage 2 of the study in participants with moderate to severe pain due to osteoarthritis in a hip and/or knee joint.

Stage 1 consists of following:

* Screening period: up to 15 days (± 2 days) (defined as Day -23 to -9)
* Washout period: 5 days (± 1 day) (defined as Day -8 to -4)
* Baseline period: 3 days (± 1 day) (defined as Day -3 to -1)
* Treatment period: 1 day (defined as Day 1): participants will be subcutaneously administered a single dose of OLP-1002 at the assigned dose level (1 μg, 3 μg, 10 μg, 25 μg, 50 μg, 80 μg)
* Follow-up period: 30 days (± 5 days) (defined as Day 2 to 30)

Approximately 30 participants will be enrolled in Stage 1 of the study

Stage 2: The study will be a double-blind, placebo-controlled, parallel-arm study of up to 2 selected single doses of OLP-1002 to evaluate the efficacy of OLP-1002 in the treatment of pain in participants with moderate to severe pain due to osteoarthritis in a knee or hip joint.

Dose levels for Stage 2 will be 1 μg and 2 μg of OLP-1002. Dose selection was based on the conclusions drawn from the internal efficacy data review analysis conducted by Sponsor from data collected in Stage 1 of the study.

Stage 2 consists of following:

* Screening Period: up to 14 days (± 2 days)
* Baseline Period: 3 days (± 1 day)
* Treatment: 1 day (± 2 days)
* Follow-up period: 42 days from last dose, D43 (± 5 days)

Approximately 90 participants will be enrolled in Stage 2 of the study

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to any study-related procedures being performed in accordance with Good Clinical Practice (GCP), International Council for Harmonisation (ICH) and local regulations.
2. Male or female aged ≥ 35 years to ≤ 70 years as of the date of enrolment into the study
3. No history of cardiac disease including arterial or venous thrombi, cardiac arrhythmia, myocardial infarction, admission to hospital for unstable angina, cardiac angioplasty or stent implantation within 90 days prior to Screening.
4. Body mass index (BMI) ≥ 18 kg/m2 < 40 kg/m2 at Screening.
5. Pain in hip or knee joints, every day for at least 1-month during the 3 months prior to Screening.

   Note: Participants must have a pain severity score of ≥ 5 based on the 3-day mean VAS score during the Baseline Period and must have recorded the pain score every day during the Baseline Period.
6. Diagnosis of Osteoarthritis (OA) of the index hip or knee: moderate to severe osteoarthritis, based on American College of Rheumatology (ACR) criteria with Kellgren Lawrence x-ray grade of at least 2, as diagnosed by the radiologist or rheumatologist.
7. Western Ontario and McMaster Universities Osteoarthritis (WOMAC) pain score of ≥ 10 out of 20 in the index hip or knee at Screening.
8. Willing and able to provide their historical use of nonsteroidal anti-inflammatory drugs (NSAIDs) either over-the-counter (OTC) per recommendation of a physician or prescribed during the past 6 months (the pain in the target knee and/or hip required).
9. Women of childbearing potential (WOCBP) must be non-pregnant and non-lactating, and must use acceptable, highly effective double contraception from Screening until 90 days after the last dose of IP. Double contraception is defined as a condom AND one other form of the following:

   1. Established hormonal contraception (for example, approved oral contraceptive pills [OCPs], long-acting implantable hormones, injectable hormones),
   2. A vaginal ring or an intrauterine device (IUD), or
   3. Documented evidence of surgical sterilisation at least 6 months prior to Screening (eg, tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women or vasectomy for men [with appropriate post-vasectomy documentation of the absence of sperm in semen] provided the male partner is a sole partner).

   Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not considered highly effective methods of birth control. A participant's treatment is acceptable.
10. Women not of childbearing potential must be postmenopausal for ≥ 12 months. Post-menopausal status will be confirmed through testing of FSH levels ≥ 40 IU/L at Screening for amenorrhoeic female participants. Female participants who are abstinent from heterosexual intercourse will also be eligible.

    Female participants who are in a same-sex relationship are not required to use contraception.
11. Male participants must be surgically sterile (>30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a WOCBP, the participant and his partner must be surgically sterile (eg, tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method from Screening until 90 days after the last dose of IP. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner that includes: OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring or an IUD.

    Male participants with a same-sex partner (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle.
12. WOCBP must have a negative pregnancy test at Screening and Day 1 and be willing to have additional pregnancy tests as required throughout the study.
13. Male participants must agree not donate sperm for at least 90 days after the last dose of IP.
14. Agree to maintain their usual levels of activity throughout the course of the study.
15. Willing to abstain from other intra-articular treatments of the joint and any joint surgery while on the study.
16. Able to comply with study procedures, including the completion of daily questionnaires.
17. Subjects suffering from moderate to severe pain secondary to diagnosed OA of the knee and/or hip joint with fit for range of age & BMI will be included with proof of COVID 19 full vaccinations and intention of the participation in the study.

Exclusion Criteria:

1. Known history or current symptomatic heart failure as per New York Heart Association (NYHA) classes II-IV, including unstable angina, myocardial infarction, serious cardiac arrhythmia, cerebral vascular accident, coronary/peripheral artery bypass graft surgery, transient ischaemic attack, or pulmonary embolism within 90 days prior to Screening.

   Participants with small pulmonary embolism not thought to put participants at higher risks of AEs may be allowed on a case-by-case basis in discussion with Sponsor.
2. History of malignancy except for basal cell carcinoma with successful removal, ALL other non-melanoma skin cancers excised successfully more than 2 years ago, and cervical intraepithelial neoplasia that has been successfully cured more than 5 years prior to the Screening Period.
3. Any of the following:

   1. Intra-articular treatment injections (including but not limited to corticosteroids, hyaluronic acid, platelet rich plasma, BOTOX®, local anaesthetics) within 3 months prior to the Screening period,
   2. QTcF > 450 ms confirmed by repeat ECG measurement,
   3. QRS duration > 120 ms confirmed by repeat ECG measurement,
   4. PR interval > 220 ms confirmed by repeat ECG measurement,
   5. Findings which would make QTc measurements difficult or QTcF data uninterpretable as per Investigator discretion,
   6. History of additional risk factors for torsades de pointes (eg, heart failure (class III/IV according to the New York Heart Association [NYHA]), hypo/hyperkalaemia, family history of long QT syndrome), or
   7. Taking any arrhythmic or arrythmia evoking agents.
4. Unable or unwilling to cease the use of all pain reducing medications and all pain reducing devices, prescription or otherwise, as of the first day of the study Baseline Period and until the End of Study visit. These include all topical and oral opioid and antiinflammatory medications, herbal and homeopathic remedies, electrostimulation therapy (EST) and neuromuscular re-education (NMRE). This excludes the use of paracetamol provided that a participant is able and willing to utilise paracetamol/acetaminophen (2 g/day) as rescue medication or up to 4 g/day for intolerable pain following consent from the PI (or designee) without prior approval from the Sponsor, as of the first day of the study, Baseline Period, and until the End of Study visit.

   Note: The participant may continue taking usual medication for maintenance of health.
5. Any of the following laboratory abnormalities within 14 days of Day 1:

   * Platelet count < 100,000 cells/mm3.
   * Total neutrophil count < 1500 cells/mm3.
   * Serum creatinine ≥ 1.5 x upper limit of normal (ULN).
   * Alanine aminotransferase (ALT) > 3.0 x ULN).
   * Aspartate aminotransferase (AST) > 3.0 x ULN.
   * Alkaline phosphatase > 2.0 x ULN.
   * Bilirubin > 1.5 x ULN.
   * Aural Temperature ≥ 38 degree Celsius or other evidence of an infection.
6. History of alcoholism, substance abuse or dependence during the 12 months prior to Screening:

   1. During the study, alcohol consumption of > 21 units per week for males and > 14 units per week for females will not be allowed. One unit of alcohol equals ½ pint (285 mL) of beer or lager, 1 glass (125 mL) of wine, or 1/6 gill (25 mL) of spirits.
   2. Positive urine drug screen (confirmed by repeat) or alcohol consumption (self-report) higher than the permissible limit, as mentioned above, at Screening or Baseline shall be excluded from the study.
7. Has an allergy or hypersensitivity to OLP-1002 or its constituents.
8. Female participants who are pregnant at Screening or are planning on becoming pregnant, or are currently breastfeeding up to 90 days from end of study.
9. Any medical condition or comorbidities as assessed by the Investigator, that could adversely impact study participation or safety, conduct of the study, or interfere with pain assessments.
10. Active skin conditions such as dermatitis, allergy, eczema, psoriasis, or abnormal skin healing. This criterion is applied in general and is not limited to the active disease at the planed injection site.
11. Tattoos, scars, or moles that in the opinion of the Investigator are likely to interfere with dosing or study assessments at any of the potential injection sites.
12. Depression of moderate or greater severity as assessed by the Investigator or via the Patient Health Questionnaire (PHQ-9 ≥10) at the Screening visit.
13. History of psychotic symptoms, whether controlled or not and/or requiring antipsychotic treatment, or history of a suicidal attempt/s within 180 days prior to Screening.
14. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndromerelated illness, acute or history of chronic hepatitis B or C. Positive tests for HIV-1 or HIV-2 antibodies, hepatitis B surface antigen, or hepatitis C antibodies at Screening.
15. Concurrent medical or arthritic conditions that could interfere with evaluation of the index joint including fibromyalgia, rheumatoid arthritis, or other inflammatory arthropathies affecting the joint eg, sciatica, diabetic neuropathy, multiple sclerosis.
16. Has undergone arthroscopic or open surgery to the joint within 180 days of Screening visit.
17. Has undergone replacement surgery of the treatment joint within 180 days of Screening visit.
18. The presence of surgical hardware /medical device or other foreign bodies in the treatment joint within 180 days of Screening visit.
19. Use or intend to use any prescription medications/products other than those medications for health conditions (eg, hypertension, diabetes or other disease), within 14 days prior to the Screening visit until the EOS (End of Study) Visit, unless deemed acceptable by the Investigator (or designee).

    Note: Prescription medication is permitted except for pain control, if deemed acceptable by the Investigator (or designee).
20. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to the Screening visit until the EOS Visit, unless deemed acceptable by the Investigator (or designee).
21. Receipt of blood products within 60 days prior to the Screening visit until the EOS Visit.
22. Donation of blood from 90 days prior to Screening until the EOS Visit, plasma from 14 days prior to Screening until the EOS Visit, or platelets from 42 days prior to Screening until the EOS Visit.
23. Poor peripheral venous access.
24. Is a Sponsor employee.
25. Has participated in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days or 5 half-lives of the IP, whichever is longer, prior to the Screening visit.
26. Has participated in any trial of a device, supplement, cognitive/behavioural therapy, physiotherapy or active exercise study within 30 days prior to the Screening visit.
27. Has previously received any dose of OLP-1002.
28. In the opinion of the Investigator (or designee), should not participate in this study.
29. Subjects who have history of or current serious illness with cardiac, vascular, cancer, infectious, mental, and laboratory abnormality will be excluded from this study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through treatment related adverse events | From baseline to end of study treatment up to 30 days
  Number of participants with treatment-related adverse events as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) criteria, v5.0.
Stage 2: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through physical examination abnormalities. | From Baseline, Day 1 (post dose), 4, 8, 15, 22, 29, 36, 43 or End of Study visit
  Any abnormalities in the body System observed by the study physician in general appearance, Ears/Eyes/Nose/Throat/Thyroid, Head, Heart, Lungs, Abdomen, Skin, Neurological, Extremities, Back, Neck, Lymph Nodes, Dentition, Nusculoskeleton.
  For example,
  1. Vital signs: out of range of normal BP systolic BP (lower than 90 and higher than 140), diastolic BP (lower than 40 and higher than 90), PR (50 -100), RR (10-20), BT(96-100 deg F)
  2. abnormal clinical exam noted by physical examining investigator.
  3. out of range of normal criteria of ECG parameters.
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through vital signs- pulse rate | From baseline to end of study treatment up to 30 days
  Measured by result of the vital signs- pulse rate
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through vital signs- blood pressure | From baseline to end of study treatment up to 30 days
  Measured by result of the Vital Sign- blood pressure (systolic and diastolic)
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through vital signs- respiratory rate | From baseline to end of study treatment up to 30 days
  Measured by result of the vital signs- respiratory rate
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through vital signs- oral aural temperature | From baseline to end of study treatment up to 30 days
  Measured by result of the vital signs- oral aural temperature
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through changes in BMI. | From screening visit, Day 1 and Day 30 or End of Study visit
  Measured by body weight in kilograms (kg) and body height (centimetres) and body weight (kilograms). BMI will be calculated by dividing the participant's body weight in kilograms by the participant's height in meters squared (kg/m2).
Stage 1: Safety of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through injection site reactions. | Stage 1: From baseline to end of study treatment up to 30 days
  The number of adverse events on injection site reaction per arms will be measured. Measured by severities or size of erythema, tenderness, bruise, and swelling will be recorded as the injection site reactions. Also, the number and rate of participants with any TEAEs will be recorded.
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through injection site reactions. | Stage 2 : From Day 1 (post dose), 4, 8, 15, 22, 29, 39, and 43 or End of Study visit
  The number of adverse events on injection site reaction per arms will be measured. Measured by severities or size of erythema, tenderness, bruise, and swelling will be recorded as the injection site reactions. Also, the number and rate of participants with any TEAEs will be recorded.
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through clinical Biochemistry results | From baseline to end of study treatment up to 30 days
  Measured by clinically significant changes in Biochemistry results
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through clinical Haematology results | From baseline to end of study treatment up to 30 days
  Measured by clinically significant changes in Haematology results
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through clinical Urinalysis results | From baseline to end of study treatment up to 30 days
  Measured by clinically significant changes in Urinalysis results
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in knee and/or hip joint through Electrocardiogram (ECG), start of atrial depolarization to start of ventricular depolarization (PR interval). | From screening visit till the end of the study visit up to 30 days
  Measured by PR interval in ECG
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Electrocardiogram (ECG) combination of the Q wave, R wave and S wave (QRS complex) | From screening Visit till the end of the study visit up to 30 days
  Measured by QRS complex result in ECG
Stage 1: Safety and tolerability of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Electrocardiogram (ECG), time from the start of the Q wave to the end of the T wave (QT interval). | From screening visit till the end of the study visit up to 30 days
  Measured by QTcF result in ECG
Stage 2: Efficacy of single dose of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through changes in Western Ontario and McMaster Osteoarthritis Index (WOMAC) | From Screening visit, Day 1 (predose), Day 4, 8, 15, 22, 29, 39 and 43 or End of Study visit
  Measured by Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale
Stage 2: Efficacy of single dose of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through changes in Visual Analogue Scale (VAS) pain score. | From Baseline, Day 1 (post dose), 4, 8, 15, 22, 29, 39 and 43 or End of Study visit
  Measured by Visual Analogue Scale (VAS) pain score

SECONDARY OUTCOMES:
Stage 1: To evaluate the efficacy of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Brief Pain Inventory questionnaire | Monitored on Day 1, 4, 8, 15, 30
  Brief Pain Inventory-Short Form (BPI-SF) is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. Patient's pain improvement will be assessed after administration of OLP-1002 on a 0 to 10 scale with 0 indicating 'no pain' and 10 indicating 'pain as worse' to assess daily pain scores.
Stage 1: To evaluate the efficacy of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Patient Global Impression of Change questionnaire (PGIC) | Monitored on Day 4, 15 and 30
  Patient's pain improvement will be evaluated based on changes in PGIC questionnaire after administration of OLP-1002 into patient with Osteoarthritis to evaluate the condition of subjects activity limitations, symptoms, emotions and overall quality of life. Patient has to chose one answer to 7 questions, each question is measured on a scale from 1 (no change/or condition has gotten worse) to 7 (condition a great deal better/considerable improvement).
Stage 1: To evaluate the efficacy of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Symptom and Quality of Life questionnaires of the KOOS. | Monitored on Day 1, 8, 15, 30
  Symptom & Quality of Life of a patient with painful Osteoarthritis will be measured by Knee Injury and Osteoarthritis Outcome Score (KOOS): For questions S1,2,3 in Symtom, using "Never (0), Rarely (1), Sometimes (2), Often (3), Always (4)" For S4,5 in Symptom, using " Always (0), Often (1), Sometimes (2), Rarely (3), Never (4)". For Quality of Life, It comes with corresponds to "Never (0), Monthly (1), Weekly (2), Daily (3), Constantly (4)" or " Not at all (0), Mildly (1), Moderately (2), Severely (3), Totally or extremely (4)".
Stage 1: To evaluate the efficacy of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Symptom and Quality of Life questionnaires of the HOOS. | Monitored on Day 8, 15, 30
  Symptom & Quality of Life of a patient with painful Osteoarthritis will be measured by Hip Injury and Osteoarthritis Outcome Score (HOOS): For Symptom, using "Never (0), Rarely (1), Sometimes (2), Often (3), Always (4)" or For Quality of Life, it comes with corresponding to "never (0), monthly (1), weekly (2), daily (3), constantly (4)" or "Not at all (0), Mild (1), Moderately (2), Severely (3), Totally or extremely (4)".
Stage 1: To evaluate the efficacy of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Western Ontario McMaster Osteoarthritis Index (WOMAC) | From baseline to end of study treatment up to Day 1, Day 4, Day 8, Day 15, Day 30
  Measured by Western Ontario and McMaster Osteoarthritis Index (WOMAC) with the pain, stiffness and physical function subscales.
  The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 4 (highest pain/ highest stiffness/ lowest function).
Stage 1: To evaluate the efficacy of OLP-1002 in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Visual Analogue Scale (VAS) | From baseline to Day 4, 8, 15 and 30
  Measured by worst daily pain intensity score on a 0 to 10 VAS scale with 0 indicating 'no pain' and 10 indicating 'pain as worse' to assess daily pain scores.
  Participants will be provided with the Patient Diary to capture daily pain intensity in a 24 hour period.
Stage 1: To evaluate maximum plasma concentration of OLP-1002 in 1 hour post administration in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint | Blood sample taken 1-hour post OLP-1002 administration on Day 1
  The previous phase 1 and 1b studies show that the practical detectable LLOQ with the currently available technique is limited to 1 nanogram/ml and LOD is 0.2 nanogram per milliter of plasma. Because of that, collecting blood samples with high dosing arms (80 mcg single dose, 160. mcg single dose, 40x5 doses, 80x5 doses) to measure OLP-1002's blood concentrating level for PK analysis method development for future OLP-1002 clincial trials. So, pK full evaluation is not available for OLP-1002 with very tiny dosing and blood concentration of OLP-1002 will be measured only in 25 mcg, 50 mcg, and 80 mcg dosing arms in stage 1.
Stage 1: Efficacy of OLP-1002 doses in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through a reduction in the use of allowed rescue pain medication | During Days 1 (postdose) to 4, Days 5 to 8, Days 9 to 15 and Days 16 to 30
  Compared with the Baseline at least a 50% reduction in the use of allowed rescue pain medication as an efficacy measure of OLP-1002 in each dose arm
Stage 2: Efficacy of OLP-1002 doses in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through a reduction in the use of allowed rescue pain medication | From baseline to Day 1 (pre dose and post dose) ,4 ,8 ,15 ,22 ,29 ,36, and 43 or Early End of Study visit
  Compared with the rescue medication usage in each dose arm at least a 50% reduction in the use of allowed rescue pain medication as an efficacy measure of OLP-1002
Stage 1: Efficacy of OLP-1002 doses in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through average use of rescue pain medication | Baseline to end of study treatment up to 30 days
  Measured by the mean (average) total dose for rescue pain medication (mg) by study day timeframe as an efficacy measure of OLP-1002 in each dose arm.
Stage 2: Efficacy of OLP-1002 doses (1 ug and 2 ug) in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through average use of rescue pain medication | From Baseline to end of study treatment up to 43 days
  Measured by the mean (average) total dose for rescue pain medication (mg) by study day timeframe as an efficacy measure of OLP-1002 in each dose arm.
Stage 1: Efficacy of OLP-1002 doses in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through average total dose for rescue pain medication (mg) by study day timeframe | Baseline to end of study treatment up to 30 days
  Measured by the average (mean) total dose for rescue pain medication (mg) by study day timeframe as an efficacy measure of OLP-1002 in each dose arm
Stage 2: Efficacy of OLP-1002 doses (1 ug and 2 ug) in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through average total dose for rescue pain medication (mg) by study day timeframe | Baseline to end of study treatment up to 43 days
  Measured by the average (mean) total dose for rescue pain medication (mg) by study day timeframe as an efficacy measure of OLP-1002 in each dose arm
Stage 1: Efficacy of OLP-1002 doses in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through time to first use of rescue pain medication | Baseline to end of study treatment up to 30 days
  Measured by the time to first use of rescue pain medication as an efficacy measure of OLP-1002 in each dose arm. It reflects the lasting period of analgesic efficacy of OLP-1002.
Stage 2: Efficacy of OLP-1002 doses (1 ug and 2 ug) in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through time to first use of rescue pain medication | Baseline to end of study treatment up to 43 days
  Measured by the time to first use of rescue pain medication as an efficacy measure of OLP-1002 in each dose arm. It reflects the lasting period of analgesic efficacy of OLP-1002.
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Treatment-related AEs and serious adverse events (SAEs) | From baseline to end of study treatment up to 43 days
  Number of participants with treatment-related adverse events as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) criteria, v5.0.
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through physical examination abnormalities. | From baseline to end of study treatment up to 43 days (on the exam dates and lab reported dates)
  Any abnormalities in the body System observed by the study physician in general appearance, Ears/Eyes/Nose/Throat/Thyroid, Head, Heart, Lungs, Abdomen, Skin, Neurological, Extremities, Back, Neck, Lymph Nodes, Dentition, Nusculoskeleton.
  For example,
  1. Vital signs: out of range of normal BP systolic BP (lower than 90 and higher than 140), diastolic BP (lower than 40 and higher than 90), PR (50 -100), RR (10-20), BT(96-100 deg F)
  2. abnormal clinical exam noted by physical examining investigator.
  3. out of range of normal criteria of ECG parameters.
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through vital signs- blood pressure | From baseline to end of study treatment up to 43 days
  Measured by result of the Vital Sign- blood pressure (systolic and diastolic)
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through vital signs- pulse rate | From baseline to end of study treatment up to 43 days
  Measured by result of the Vital Sign- pulse rate
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through vital signs- respiratory rate | From baseline to end of study treatment up to 43 days
  Measured by result of the Vital Sign-respiratory rate
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through vital signs- oral aural temperature | From baseline to end of study treatment up to 43 days
  Measured by result of the Vital Sign- oral aural temperature
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through injection site reactions. | From baseline to end of study treatment up to 43 days
  Measured by result of adverse events recorded as injection site reactions
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in knee and/or hip through changes in BMI. | From screening visit till the end of the study visit up to 43 days
  Measured by body weight in kilograms (kg) and body height (centimetres) and body weight (kilograms). BMI will be calculated by dividing the participant's body weight in kilograms by the participant's height in meters squared (kg/m2).
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in knee and/or hip joint through through Electrocardiogram (ECG), combination of the Q wave, R wave and S wave (QRS complex) | From screening visit till the end of the study visit up to 43 days
  Measured by QRS interval in ECG
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in knee and/or hip joint through ECG, start of atrial depolarization to start of ventricular depolarization (PR interval) | From screening visit till the end of the study visit up to 43 days
  Measured by PR interval in ECG
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Electrocardiogram (ECG), time from start of Q wave to end of T wave (QT interval). | From screening visit till the end of the study visit up to 43 days
  Measured by QTcF result in ECG
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through clinical Biochemistry results | From baseline to end of study visit up to 43 days
  Measured by clinically significant changes in Biochemistry results from previous results and out of range of laboratory results for the safety issue. There is no biomarker up to now for the evaluation of the pain reduction unfortunately. The clinical Biochemistry includes AST(U/L), ALT (U/L), GGT (IU/L), ALP (U/L), creatine kinase (U/L), amylase (U/L), serum lipase (U/L), total bilirubin (umol/L), blood urea nitrogen (mg/dL), creatine (umol/L), eGFR (mL/min/1.7 3m^2), uric acid (mmol/L), albumin (g/L), urine albumin/creatinine ratio (ug/mg Cr), total protein (g/L), glucose (mmol/L), cholesterol (mg/dL), triglycerides (mmol/L), potassium (mmol/L), sodium (mmol/L), calcium (mmol/L).
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through clinical hematology results | From baseline to end of study visit up to 43 days
  Measured by clinically significant changes in hematology results from previous results and out of range of laboratory results for the safety issue. Clinical hematology includes hemoglobin(g/L), hematocrit (%), red blood cell count (10^12/L), erythrocyte sedimentation rate (mm/hr), mean cell hemoglobin (pg), mean cell volume(fL), mean cell hemoglobin concentration (g/L), white blood cell count (10^9/L), platelet blood count (10^9/L), and differential blood count (automated).
Stage 2: Safety of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through clinical urinalysis | From baseline to end of study visit up to 43 days
  Measured by clinically significant changes in urinalysis results from previous results and out of range of laboratory results for the safety issue. The clinical urinalysis includes nitrites (negative), leukocytes (WBCs/uL), protein (mg/dL), glucose (mg/dL), ketones (mg/dl), blood (RBCs/uL), negative common logarithm of hydrogen ion concentration (pH), specific gravity (1.005 ~1.030), creatinine (mmoL), bilirubin (mg/dL), and urobilinogen (mg/dL).
Stage 2: Efficacy of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through reduction in use of allowed rescue pain medication | During Days 1 (postdose) to 4, Days 5 to 8, Days 9 to 15, Days 16 to 22, Days 23 to 29, Days 30 to 36 and Days 37 to 43.
  Compared with Baseline at least 50% reduction in use of allowed rescue pain medication
Stage 2: Efficacy of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through change in KOOS Symptoms and QoL Subscale | On Days 8, 15, 22, 29, 36 and 43 after administration of OLP-1002.
  Change from Baseline in KOOS Symptoms and QoL Subscale: For Symtpom questions S1,2,3, using "Never (0), Rarely (1), Sometimes (2), Often (3), Always (4)" or S4,5 " Always (0), Often (1), Sometimes (2), Rarely (3), Never (4). For QoL comes with corresponding to " Never (0), Monthly (1), Daily (3), Constantly (4)" or Not at all (0), Mildly (1), Moderate (2), Severely (3), Totally or extremely (4)".
Stage 2: Efficacy of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through change in HOOS Symptoms and QoL Subscale | On Days 8, 15, 22, 29, 36 and end of study visit day 43 after administration of OLP-1002.
  Change from Baseline in HOOS Symptoms and QoL Subscale: For Symptom question S1,2,3 using "Never (0), Rarely (1), Sometimes (2), Often (3), Always (4)". For Quality of Life comes with corresponding to " Never (0), Monthly (1), Weekly (2), Daily (3), Constantly (4)" or "Not at all (0), Mildly (1), Moderately (2), Severely (3), Totally or extremely (4)" for severity
Stage 2: Efficacy of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Brief Pain Inventory questionnaire | Days 4, 8, 15, 22, 29, 36 and end of study visit day 43 after administration of OLP-1002.
  Brief Pain Inventory-Short Form (BPI-SF) is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. Patient's pain improvement will be assessed after administration of OLP-1002 on a 0 to 10 scale with 0 indicating 'no pain' and 10 indicating 'pain as worse' to assess daily pain scores.
Stage 2: Efficacy of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through Patient Global Impression of Change questionnaire (PGIC) | Days 4, 15, 22, 29, 36, and end of study visit day 43 after administration of OLP-1002.
  Patient's pain improvement will be evaluated based on changes in PGIC questionnaire after administration of OLP-1002 into patient with Osteoarthritis to evaluate the condition of subjects activity limitations, symptoms, emotions and overall quality of life. Patient has to chose one answer to 7 questions, each question is measured on a scale from 1 (no change/or condition has gotten worse) to 7 (condition a great deal better/considerable improvement).
Stage 2: Efficacy of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through changes in Western Ontario and McMaster Osteoarthritis Index (WOMAC) | Days 4, 8, 15, 22, 29, 36 and end of study visit day 43 after administration of OLP-1002.
  Measured by Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale
Stage 2: Efficacy of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through changes in Visual Analogue Scale (VAS) | Baseline to end of study visit day 43 after administration of OLP-1002.
  Measured by worst daily pain intensity score on a 0 to 10 VAS scale with 0 indicating 'no pain' and 10 indicating 'pain as worse' to assess daily pain scores.
  Participants will be provided with the Patient Diary to capture daily pain intensity in a 24 hour period.
Stage 2: Efficacy of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through changes in the use of rescue pain medication | Baseline to end of study visit day 43 after administration of OLP-1002.
  Measured by rescue pain medication use by study day timeframe
Stage 2: Efficacy of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through average use of rescue pain medication | Baseline to end of study visit day 43 after administration of OLP-1002.
  Measured by the mean (average) total dose for rescue pain medication (mg) by study day timeframe.
Stage 2: Efficacy of OLP-1002 (1μg and 2μg) compared to placebo in adults with moderate to severe pain due to osteoarthritis in a knee and/or hip joint through time to first use of rescue pain medication | Baseline to end of study visit day 43 after administration of OLP-1002.
  Measured by the time to first use of rescue pain medication

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ostor, Principal Investigator — Emeritus Research
Locations (7):
- Australia (7):
  - Northern Beaches Clinical Research, Brookvale, New South Wales
  - Novatrials, Kotara, New South Wales
  - Sutherland Shire Clinical Research, Miranda, New South Wales
  - Emeritus Research, Sydney, New South Wales
  - AusTrials, Taringa, Queensland
  - AusTrials, Wellers Hill, Queensland
  - Emeritus Research, Melbourne, Victoria